CLINICAL TRIAL: NCT05286164
Title: Eltrombopag Treatment and Analysis of Bone Marrow Environment in Patients With Prolonged Bone Marrow Toxicity After CART Treatment
Brief Title: Eltrombopag Treatment in Patients With Prolonged BM Toxicity After CART
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0248-21
Record Dates: First submitted 2022-02-24; First posted 2022-03-18 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-03

CONDITIONS: CART Treatment; B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — eltrombopag

STUDY DESIGN:
Intervention Model Description: Patients with bone marrow aplasia for more than 3 weeks after CART administration will receive eltrombopag treatment at a dose of 150 mg for 8 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eltrombopag (Experimental): Patients with bone marrow aplasia for more than 30 days after CART treatment
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — Eltrombopag 150 mg QD for 8 weeks

SUMMARY:
Treatment with chimeric antigen receptor-T cell (CAR-T) is successful in patients who have not responded to chemotherapy or bone marrow transplantation but it may provoke side effects and long-term complications. Early and specific side effects include cytokine release syndrome and neurological toxicity. In addition, there are also late side effects. The most prominent of which is bone marrow damage and lack of recovery of blood counts after treatment.

In this study, patients with prolong aplasia after CAR-T will recieve eltrombopag to enahnce bone marrow recovery.

DETAILED DESCRIPTION:
CAR-T therapy is the standrad of care in patients with relapse/refractory B cell agressive lymphoproliferative diseases. Prolonged cytopenia is a not uncommon side effect and is associated with susbstantial morbidity and in severe cases also with mortality. The pathobiologic process that causes bone marrow injury is not known and in order to find appropriate treatment it is important to expand the knowledge regarding this toxicity. Current treatment options for bone marrow suppression includes growth factor therapy (GCSF), steroids and immunoglobulins. .

The investigators hypothesize that CART cells directly suppress or create inflammatory process in bone marrow. This process may resemble aplastic anemia, a marrow aplasia that occurs secondary to inflammatory process.

Treatment of aplastic anemia is based on the administration of eltrombopag, that causes a thrombopoietin-mimetic blood cells to develop and multiply. This treatment demonstrated an increase in the amount of platelets and neutrophils in patients with aplastic anemia and is approved by the health authorities around the world and in Israel as a standard treatment for this disease. There are several reports of successful use of altrombopag in patients after CART who have developed marrow toxicity and in patients after bone marrow transplantation whose blood counts are low.

In this study, patients with prologed aplasia after CART cells therapy, will be given eltrombopag in a purpose to incrase bone marrow function. In addition, the investigators will perform several assays to shed more light on the basic pathologic process that causes the bone marrow aplasia.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate in the study and able to sign an informed consent form.
2. Patients with B cell lymphoma or multiple myeloma who were treated with CART and demonstrated cytopenia on day 14 after CART administration. Cytopenia definition: absolute neutrophil count <500 neutrophils/ul and/or platelets <50,000 mm3
3. Bone marrow demonstrates hypoplasia (cellularity less than 30%) 14 days after CART administration.

   -

Exclusion Criteria:

1. Creatine > 2.5 mg / dL
2. Disorder in liver enzymes: bilirubin above 2 mg/dl , AST or ALT 5 times the normal.
3. Active infection
4. Active hemophagocytic syndrome
5. Evidence of a viral or pharmacological disease that causes bone marrow injury
6. Susceptibility to eltrombopag
7. Evidence of disease in the bone marrow -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
The percentage of cellularity | up to 12 weeks (4 weeks from CART treatment and additional 8 weeks of treatment with eltrombopag)
  Efficacy of eltrombopag treatment will be measured based on recovery of blood counts and recovery of bone marrow aplasia (measured as percentage of cellularity)
Identify the mechanism for the appearance of late bone marrow toxicity | 12 weeks from CART treatment
  Identification of the mechanism for the CART- associated bone marrow aplasia will be based on cytokines profile, T cell subclasses analyses and single cell RNA sequencing. This will enable the investigators to shed more light on the pathologic process that connects CART cells admisnitration and bone marrow apasia.

CONTACTS AND LOCATIONS:
Overall Officials: Ron Ram, Prof., Principal Investigator — Sourasky Medical Center
Locations (1):
- Tel-Aviv Sourasky Medicak center / BMT Unit, Tel Aviv, Israel